CLINICAL TRIAL: NCT06878066
Title: The Efficacy and Safety of Intravenous Thrombolysis in Acute Ischemic Stroke Patients With Recent Ingestion of Factor Xa-inhibitors Trial (SIFT)
Brief Title: Thrombolysis in Factor Xa-inhibitors Trial
Acronym: SIFT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guri Hagberg (Other)
Collaborators: Klinbeforsk (Other); Clinical Trial Unit (CTU), Oslo University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Guri Hagberg, MD, PhD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-509907-34-01; 2023-509907-34-01 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Stroke (in Patients With Atrial Fibrillation); Ischemic Stroke; Acute Ischemic Stroke; Anticoagulant Therapy; Factor Xa Inhibitor; Intracranial Hemorrhages; Hemorrhagic Transformation Due to Acute Stroke; Bleeding in the Brain
Keywords: Thrombolysis; Acute Ischemic Stroke; Ischemic Stroke; Factor Xa Inhibitors; Atrial Fibrillation-Related Stroke; Intravenous Thrombolysis; Tissue Plasminogen Activator; Tenecteplase; Alteplase; Symptomatic Intracranial Hemorrhage; SIFT Trial; Stroke; Acute stroke; Direct Oral Anticoagulants; DOACs
MeSH Terms: conditions — Stroke; Ischemic Stroke; Intracranial Hemorrhages | interventions — Thrombolytic Therapy; Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Intervention Model Description: A pragmatic phase III, multicenter, prospective, randomized, open label, blinded endpoint (PROBE), registry-linked, trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVT (Active Comparator): Intravenous Thrombolysis (IVT) with Alteplase or Tenecteplase
  Interventions: Drug: thrombolysis therapy
- NO IVT (No Intervention): Standard Care Without Thrombolysis

INTERVENTIONS:
Drug: thrombolysis therapy — All treatment and monitoring routines are according to the hospitals' standard operating procedures (SOP), and both drugs (Alteplase (ALP) and Tenecteplase (TNK)) are approved drugs for the indication AIS with similar efficacy and safety profile. SIFT is designed to test the hypothesis that intravenous thrombolysis (IVT) (tenecteplase 0.25 mg/kg or alteplase 0.9 mg/kg intravenously) is efficient and safe in acute ischemic stroke patients (AIS) with recent ingestion (last 48 hours) of an Factor Xa (FXa) inhibitor who otherwise are eligible for IVT.
  Other Names: Alteplase; Tenecteplase
  Arms: IVT

SUMMARY:
This study looks at whether stroke patients who take FXa inhibitors (a type of blood thinner) can safely receive clot-busting treatment (IVT). IVT is a common emergency treatment for stroke, but current guidelines say it should not be given to people who have taken FXa inhibitors in the last 48 hours. This is because doctors worry that IVT might cause dangerous bleeding in the brain.

However, new research suggests that IVT might be safe for these patients. Some studies even show that stroke patients on FXa inhibitors who receive IVT do not have a higher risk of brain bleeding than other stroke patients. But because these studies were not designed as full medical trials, doctors still avoid IVT for this group.

The SIFT trial will compare two groups of stroke patients who take FXa inhibitors:

One group will receive IVT to see if it helps them recover better. One group will not receive IVT, which is the current standard. Doctors will check if IVT helps with recovery and if it causes any serious bleeding. If IVT is found to be safe and effective, this study could change stroke treatment guidelines and help more patients get life-saving care.

Right now, some guidelines say that stroke patients on FXa inhibitors should have a blood test before getting IVT, to measure how much of the drug is in their system. But these tests are not available in most hospitals, and waiting for results could delay important treatment. The SIFT trial will not require this test before giving IVT.

More and more people use FXa inhibitors to prevent strokes, but right now, they are being denied IVT based on old rules. If this study proves that IVT is safe for them, it could help doctors give better care to thousands of stroke patients.

DETAILED DESCRIPTION:
The SIFT trial is a pragmatic phase III, multicenter, prospective, randomized, open-label, blinded-endpoint (PROBE), registry-linked trial. It is designed to test the hypothesis that intravenous thrombolysis (IVT) is both safe and effective in patients with acute ischemic stroke (AIS) who have ingested a Factor Xa (FXa) inhibitor within the last 48 hours and are otherwise eligible for IVT. The study aims to address the current limitations in stroke guidelines, which recommend against IVT in these patients due to concerns of symptomatic intracranial hemorrhage (sICH). However, these recommendations are based on data from vitamin K antagonist (VKA) studies rather than direct evidence from randomized clinical trials (RCTs) involving FXa inhibitors. Observational data suggest that IVT in patients on FXa inhibitors is safe and effective, but a well-monitored RCT is necessary to confirm these findings.

All treatment and monitoring routines in the study follow hospital standard operating procedures (SOPs), and both alteplase (ALP) and tenecteplase (TNK) are approved drugs for AIS, with similar efficacy and safety profiles. IVT is known to be an effective treatment for disabling AIS, improving functional outcomes when administered within 4.5 hours of symptom onset. FXa inhibitors have largely replaced warfarin due to their better safety profile, reducing the risk of hemorrhagic complications by 50% compared to VKAs. The concern over sICH remains a major reason why patients on FXa inhibitors are often excluded from IVT, yet research suggests that the net benefit of IVT outweighs the risks, even with an sICH rate of up to 8%.

The primary objective of the study is to compare early neurological improvement (ENI) in patients treated with IVT versus those receiving standard care. Secondary objectives include assessing clinical neurological improvement, infarct volume changes on imaging, functional outcomes, rates of sICH, any intracranial hemorrhage (ICH) after IVT, and overall mortality. The study has a planned recruitment of 300 patients, with a 2:1 allocation favoring IVT. The sample size is designed to provide sufficient power for primary and secondary analyses, including the safety assessment of sICH rates. The study will be conducted across emergency departments and acute stroke units in Norway.

Eligibility criteria include patients aged 18 or older who have ingested an FXa inhibitor within 48 hours before symptom onset (or have an ongoing prescription if the exact timing of last ingestion is unknown). Patients must have a clinical diagnosis of AIS with disabling neurological deficits and present within 4.5 hours of symptom onset or after awakening with symptoms, confirmed by imaging. Informed consent is required. Patients with contraindications to alteplase or tenecteplase, those planned for endovascular treatment due to isolated large vessel occlusion (LVO) in the internal carotid artery (ICA) or middle cerebral artery (MCA) with expected rapid intervention, those using dabigatran, or those deemed at high risk by their treating physician are excluded.

Participants randomized to the IVT arm will receive either alteplase (0.9 mg/kg with a 10% bolus and 90% infusion over 60 minutes) or tenecteplase (0.25 mg/kg single bolus) according to local SOPs. The control group will receive 300 mg of aspirin and no IVT, in line with current practice guidelines. The study duration is planned from 2025 to 2029, with termination by December 2030 unless safety concerns necessitate earlier closure. The estimated duration of patient follow-up is 90 days.

The study follows an open-label, blinded-endpoint design, with patient randomization handled via a computerized system (Viedoc). Randomization is stratified by age and baseline NIH Stroke Scale (NIHSS) score. The primary outcome measure is early neurological improvement, defined as an NIHSS reduction of ≥8 points or an NIHSS score of 0-1 at 24 hours. Secondary outcomes include percentage change in NIHSS from baseline, infarct volume at 24 hours, functional outcomes at 90 days, and the incidence of sICH and any ICH within 36 hours. Death within 90 days is also assessed.

The primary analysis will use a logistic regression model, adjusting for age, NIHSS score, and time to treatment. Safety monitoring will be continuous, with an early stopping mechanism in place if the sICH rate in the IVT arm is deemed unacceptably high. The study's impact could be substantial; if IVT is proven safe and effective in AIS patients on FXa inhibitors, it would significantly influence stroke management, enabling more patients to receive IVT and reducing post-stroke disability. These findings would contribute to international discussions and could lead to guideline changes worldwide, allowing all IVT-capable centers to offer immediate, effective treatment to a growing patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age or older.
2. Ingestion of FXa inhibitors within the last 48 hours of symptom onset (or ongoing prescription of FXa inhibitor if unknown)
3. Clinical diagnosis of AIS with disabling neurological deficit
4. Presenting within 4.5 h of symptom onset or after awakening with symptoms of AIS with FLAIR-DWI mismatch on MRI as judged by the (neuro-) radiologist.
5. Informed consent

Exclusion Criteria:

1. Endovascular treatment eligible patients with isolated large vessel occlusion of the intracranial internal carotid artery (ICA), the M1 segment of the middle cerebral artery (MCA), or both confirmed by CT or MR angiography and expected time from randomization to groin puncture of <30 minutes.
2. Systolic BP >185 mmHg or diastolic BP >110 mmHg despite antihypertensive treatment.
3. Known bleeding diathesis; manifest or recent severe bleeding; significant bleeding disorder last 6 months.
4. Arterial puncture at a non-compressible site; biopsy or lumbar puncture <7 days; major surgery, traumatic external heart massage, obstetrical delivery or serious trauma <14 days; history of intracranial haemorrhage; stroke <2 months, CNS neurosurgery <2 months; serious head trauma <2 months; pericarditis; sepsis; bacterial endocarditis; pericarditis; acute pancreatitis; neoplasm with increased bleeding risk; any serious medical illness likely to interact with treatment (i.e. aortic dissection); confounding pre-existent neurological or psychiatric disease.
5. Any condition that, in the opinion of the treating physician, puts a patient at risk if treated with thrombolysis (i.e. signs of cerebral hemorrhage, known cerebral amyloid angiopathy, CT with signs of early ischemia greater than one-third of the middle cerebral artery territory).

   Prior/Concomitant Therapy
6. Use of a) direct thrombin (II) inhibitor (Dabigatran) or b) warfarin with an INR ≥1.8; c) heparin <48 h; d) treatment dose of LMWH <24 h.

   Prior/Concurrent Clinical Study Experience
7. Hypersensitivity to Alteplase or Tenecteplase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Early neurological improvement (ENI) | 24 hours (22-36 h).
  Early neurological improvement, defined as a reduction of ≥8 points on the National Institutes of Health Stroke Scale (NIHSS), or NIHSS of 0-1 at 24 hours (22-36 h).

SECONDARY OUTCOMES:
NIHSS change | 24 hours (22-36 hours)
  Percentage change in NIHSS (National Institutes of Health Stroke Scale) from baseline to 24 hours (22-36 hours).
  To compare clinical neurological improvement between patients treated with IVT and patients treated with the current standard of care.
  The National Institutes of Health Stroke Scale (NIHSS) consists of 11 items, each assessing a distinct neurological function, with scores ranging from 0 to 4. A score of 0 typically reflects normal function for the given domain, while higher scores indicate varying degrees of impairment. The total NIHSS score is derived by summing the individual item scores, with the total score representing the overall severity of neurological deficit. The scale's total score ranges from 0 to 42, where 0 indicates no neurological impairment, and 42 signifies the most severe impairment.
Infarct volume | 24 hours ± 12 hours.
  Percent change in infarct volume at 24 hours ± 12 hours. To compare infarct volume on CT/MRI (computed tomography/magnetic resonance imaging) at 24 hours ±12 hours between patients treated with intravenous thrombolysis and patients treated with the current standard of care, infarct volume is defined as follows: For magnetic resonance imaging, infarct volume is a visible hyperintense area on both T2 FLAIR (T2 Fluid-Attenuated Inversion Recovery) and diffusion-weighted imaging (DWI) with a decrease in apparent diffusion coefficient (ADC). For computed tomography, infarct volume involves manual delineation of the hypodense infarct area.
mRS (modified Rankin Scale) score | 90 days (+/- 2 weeks)
  Obtaining a good functional outcome (mRS 0-2) at day 90 (+/- 2weeks); obtaining an excellent functional outcome (mRS 0-1) at day 90 (+/- 2 weeks); mRS category at day 90 (+/- 2 weeks).
  To compare functional outcome between patients treated with IVT and patients treated with the current standard of care.
  The Modified Rankin Scale (MRS) assesses the degree of disability or dependence in daily activities following a stroke or other neurological event. It ranges from 0, indicating no symptoms, to 6, indicating death. The scale measures levels of disability from no impairment (0) to severe disability requiring constant care (5), with intermediate levels reflecting varying degrees of functional limitation and need for assistance.
Symptomatic Intracranial Hemorrhage (sICH) | 36 hours
  Occurrence of sICH on CT/MRI within 36 hours post IVT causally related to an increase of 4 points or more on the NIHSS.
  To compare the rate of sICH in AIS patient with ingestion of FXa inhibitors within the last 48 hours and treated with IVT within 4.5 hours after stroke onset versus the expected sICH rate seen in Norway in patients not taking FXa inhibitors prior to IVT.
Any Intracranial Hemorrhage (ICH) | 36 hours
  The rate of any ICH in the treatment arm on CT/MR within 36 hours post IVT.
Death | 90 days
  To compare the number of deaths of participants between patients treated with IVT and patients treated with the current standard of care, within 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Ihle-Hansen, MD, PhD, Principal Investigator — Dept. of Medicine, Baerum Hospital
Locations (13):
- Norway (13):
  - Dept. of Medicine, Baerum Hospital, Bærum, Gjettum
  - Dept of Medicine, Helse More and Romsdal Health Trust, Aalesund Hospital, Ålesund
  - Dept of Medicine, Haraldsplass deaconal Hospital, Bergen
  - Dept. Of Neurology, Haukeland University Hopsital, Bergen
  - Dept of Neurology, Drammen Hospital Trust, Drammen
  - Dept of Neurology, Ostfold Hospital Trust, Kalnes, Grålum
  - Dept of Neurology, Hospital of Southern Norway, SSHF, Kristiansand
  - Dept of Neurology, Innlandet Hospital Trust, Lillehammer, Lillehammer
  - Dept. of Neurology, Oslo University Hospital, Oslo
  - Dept of Neurology, Stavanger University Hospital, Stavanger
  - Dept. of Neurology, Tromso University Hospital, Tromsø
  - Dept. Of Medicine, St.Olav Hospital, Trondheim, Trondheim
  - Dept of Neurology, Vesfold Hospital Trust, Tonsberg, Tønsberg

REFERENCES:
- See also: CTIS Portal where the primary trial protocol and references are accessible — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-509907-34-01